CLINICAL TRIAL: NCT01412554
Title: Impact of INsulin Sensitivity on Cardiovascular Risk Markers During 10-20 Years of FOllow-up
Brief Title: Impact of INsulin Sensitivity on Cardiovascular Risk Markers During 10-20 Years of FOllow up
Acronym: INFO
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Tonje Amb Aksnes, PhD, Oslo University Hospital
Other Study IDs: 2010/3339
Record Dates: First submitted 2011-07-22; First posted 2011-08-09 (Estimated); Results first posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-09

CONDITIONS: Diabetes Mellitus; Hypertension; Ischemic Heart Disease; Stroke
Keywords: Insulin resistance; Diabetes mellitus; Adipositas
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Myocardial Ischemia; Stroke; Insulin Resistance; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — whole blood, serum, white cells, urine, fat tissue cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Longitudinal Insulin Sensitivity: The participants were examined using the hyperinsulinaemic isoglycaemic glucose clamp technique which is the gold standard to assess insulin sensitivity.

SUMMARY:
The purpose of this study is to identify risk factors for insulin resistance and to investigate the influence of insulin sensitivity on development of cardiovascular risk markers like blood pressure, heart rate, body build (weight, BMI, waist-hip ratio, skinfold thickness), reduced insulin sensitivity, diabetes mellitus, dyslipidaemia, and sympathoadrenal activity or manifest cardiovascular disease among young men during 10-20 years.

DETAILED DESCRIPTION:
In 1988 Reaven described a syndrome designed "syndrome X" based on the clustering of resistance to insulin-stimulated glucose uptake, hyperinsulinaemia, hyperglycaemia, increased triglycerides, decreased high-density lipoprotein (HDL) cholesterol and high blood pressure and proposed insulin resistance as the common feature and the aetiology of the syndrome. Later obesity and the sympathetic nervous system have been proposed as pathogenic factors of the metabolic syndrome, and still major controversy exists regarding its precise aetiology and different definitions of metabolic syndrome are also discussed.

Insulin resistance is a growing epidemic concern in both industrialized and developing countries. It is one of the components of the metabolic syndrome, and plays an important role in the pathogenesis of type 2 diabetes. In view of the predicted increase in the number of diabetic patients during the coming decades, further information about risk factors and pathophysiology of diabetes are of utmost importance for early detection and possible prevention and early treatment from both a medical and a financial perspective. Our research group has for decades studied the pathophysiology of insulin resistance, hypertension, sympathoadrenal hyperreactivity and dyslipidaemia. We have also recently finished a long-term follow up study of subjects based on their cardiovascular and sympathetic responses to mental stress.

During 1991-2002 healthy young men recruited from the military enlistments in the Oslo/Akershus area were examined at Center of Cardiovascular and Renal Research, Division of Medicine, Oslo University Hospital, Ullevål. Young, healthy men, mean age of 21, were examined using the hyperinsulinaemic isoglycaemic glucose clamp technique, which is the gold standard to assess insulin sensitivity. The present study aims to re-examine these subjects in order to investigate the influence of insulin sensitivity on development of cardiovascular risk factors and diabetes. We therefore have a unique opportunity to perform a true, long-term follow-up study of a homogenous sample of subjects of same race and gender which may provide new insights into various pathophysiological mechanisms in diabetes and cardiovascular disease including elucidating the connections between insulin resistance, changes in parameters of body build, blood pressure and sympathetic over-activity. Clarifying these mechanisms are of direct importance for the entire population. There has to our knowledge not been any previous long-term follow-up on subjects based on their insulin resistance measured with this gold standard technique.

We now want to re-examine the same subject to investigate the influence of insulin sensitivity on development of cardiovascular risk factors like blood pressure, heart rate, body build (weight, BMI, waist-hip ration, skinfold thickness), reduced insulin sensitivity, diabetes mellitus, dyslipidaemia, and sympathoadrenal activity or manifest cardiovascular disease among young men during 10-20 years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Completed hyperinsulinemic glucose clamp

Exclusion Criteria:

* Missing agreement
* No contact information

Ages: 30 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 103 men previously examined with hyperinsulinemic glucose clamp, measuring insulin sensitivity, at Center of Cardiovascular and Renal Research, Division of Medicine, Oslo University Hospital, Ullevål.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2011-08; Primary Completion 2014-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sverre E Kjeldsen, PhD, Study Director — Oslo Univeristy Hospital
Locations (1):
- Section of Cardiovascular and Renal Research, Oslo, Norway

REFERENCES:
- [Derived] Akra S, Aksnes TA, Flaa A, Eggesbo HB, Opstad TB, Njerve IU, Seljeflot I. Markers of remodeling in subcutaneous adipose tissue are strongly associated with overweight and insulin sensitivity in healthy non-obese men. Sci Rep. 2020 Aug 20;10(1):14055. doi: 10.1038/s41598-020-71109-4. PMID 32820223
- [Derived] Skarn SN, Eggesbo HB, Flaa A, Kjeldsen SE, Rostrup M, Brunborg C, Reims HM, Aksnes TA. Predictors of abdominal adipose tissue compartments: 18-year follow-up of young men with and without family history of diabetes. Eur J Intern Med. 2016 Apr;29:26-31. doi: 10.1016/j.ejim.2015.11.027. Epub 2015 Dec 23. PMID 26712453
- See also: Homepage for Section of Cardiovascular and Renal Research — https://www.med.uio.no/klinmed/english/research/groups/cardiovascular-and-renal/index.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During 1991-96 men from the military enlistments were examined at Center of Cardiovascular and Renal Research, Division of Medicine, Oslo University Hospital, Ullevål, using hyperinsulinaemic isoglycaemic glucose clamp technique to assess insulin sensitivity.
  They were re-invited to participate in the presented study during 2012-13.
Pre-assignment Details: 103 consented to participation.
Period: Overall Study
Arm/Group | Longitudinal Insulin Sensitivity
Started | 103 (103 persons re-examined in 2012-13 out of 158 persons originally examined in 1991-96.)
Completed | 103
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Longitudinal Insulin Sensitivity
Number analyzed (Participants) | 103
Age, Continuous [Median (Standard Deviation); unit: years] | 40 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 103

OUTCOME MEASURES:

1. Primary Outcome: Exploring Insulin Sensitivity After 10-20 Years of Follow-up
Description: The primary outcome is insulin sensitivity measured as the glucose disposal rate (GDR) (mg/kg/min), calculated from the average glucose infusion rate during the last 20 minutes of a 120 minutes hyperinsulinaemic isoglycaemic glucose clamp.
Time Frame: One-day visit and the analyses will be done when all patients are examined in the period 2012-2013
Measure: Mean (Standard Deviation); unit: mg/kg/min
Arm/Group | Longitudinal Insulin Sensitivity
Number analyzed (Participants) | 103
mg/kg/min | 7 (2)
Statistical Analysis 1: Comparison: Longitudinal Insulin Sensitivity; Only an observational follow-up study; Test type: Other — Only descriptive statistics; p < 0.05, Spearman; The degree of tracking was assessed by Spearman's rank or Pearson's correlation coefficient; The degree of tracking was assessed by Spearman's rank or Pearson's correlation coefficient

2. Primary Outcome: Exploring Insulin Sensitivity After 10-20 Years of Follow-up
Description: as for outcome 1
Time Frame: 20 years
Reporting Status: Not Posted

3. Secondary Outcome: Sympathoadrenal Activity During Rest and Stress Tests
Description: A mental arithmetic stress test will be announced and performed immediately after the glucose clamp, to assess the effects of increased adrenaline and noradrenaline when hepatic glucose production is suppressed by hyperinsulinaemia. Blood pressure, heart rate and catecholamine blood-levels are measured at pre-defined intervals.
Time Frame: One-day visit and analyses will be done during 2012-2013
Reporting Status: Not Posted

4. Secondary Outcome: Echocardiography
Description: Transthoracic echocardiography will be performed using a VIVID E9 (or VIVID 7) echocardiographic scanner (GE Vingmed, Horten) with 1,7-MHz probe in second harmonic mode and optimal gain and contrast.Left ventricular (LV) internal dimension, intraventricular septal thickness and LV posterior wall thickness will be measured as well as epicardial adipose tissue. We will also evaluate biplane Simpson ejection fraction and valvular incompetence
Time Frame: One-day visit, final analyses 2012-2013
Reporting Status: Not Posted

5. Secondary Outcome: Ultrasound Abdomen
Description: Ultrasound quantification of abdominal adipose tissue
Time Frame: One-day visit. Final analyses of the whole cohort during 2012-2013
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 month
Description: No adverse evnts
Arm/Group | Longitudinal Insulin Sensitivity
All-Cause Mortality (participants affected / at risk) | 0/103
Serious Adverse Events (participants affected / at risk) | 0/103
Other Adverse Events (participants affected / at risk) | 0/103

LIMITATIONS AND CAVEATS:
Results limited to the study group

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No